CLINICAL TRIAL: NCT04208425
Title: Promoting Resilience in Teens With ASD
Acronym: PRITA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Collaborators: Society of Clinical Child & Adolescent Psychology (Unknown); Autism Research Institute (Unknown)
Responsible Party: Principal Investigator, Matthew Daniel Lerner, Associate Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2019-00280; AWD00001042 (Other Grant/Funding Number: Society of Clinical Child & Adolescent Psychology); AWD00001244 (Other Grant/Funding Number: Autism Research Institute)
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Anxiety; Depression; Autism; Autism Spectrum Disorder; Single Session Intervention; ASD; SSI
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Depression; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This study will be a two-arm randomized controlled trial, including one active intervention conditions and one active control condition. Adolescents (and one caregiver per adolescent participant) will visit the Social Competence and Treatment Lab in the Department of Psychology at Stony Brook University. This lab visit will last approximately 2.5 hours. Adolescents and parents will complete baseline questionnaires (see sections below for details). Participants will then be randomized to one of two intervention conditions, using Qualtrics built in functionality: the single session growth mindset intervention (SSI GMI), or an active control program, designed to replicate supportive therapy (ST) and tested in previous work. Immediately after intervention completion, adolescents will complete a brief post-intervention questionnaire battery. Adolescents and parents will then be asked to complete online follow-up questionnaire batteries 3-months post-intervention.
Who Masked: Participant, Investigator
Masking Description: Participants in the study will be masked by using Qualtrics built in randomization function.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Personality (Experimental): The web-based growth mindset intervention, called Project Personality, is delivered entirely via Qualtrics and takes approximately 30 minutes to complete. All intervention activities are self-administered by youth and delivered in a web-based format, including illustrations and audio-recordings of text. Intervention content is designed to maximize relevance for youths experiencing symptoms of depression, including excessive sadness and hopelessness.
  Interventions: Behavioral: Project Personality
- Sharing Feelings Intervention (Active Comparator): The Sharing Feelings Intervention is delivered entirely via Qualtrics, is self-administered by youth, and takes approximately 30 minutes to complete. It is structurally similar to the growth mindset intervention, but it is designed to mimic supportive therapy (ST). The goals of the ST intervention is to encourage youths to identify and express feelings to close others; the intervention does not teach or emphasize specific skills or beliefs. In previous clinical trials, ST has resulted in significantly fewer reductions in youth internalizing problems compared to cognitive-behavioral and growth mindset interventions.
  Interventions: Behavioral: Sharing Feelings Intervention

INTERVENTIONS:
Behavioral: Project Personality — The intervention includes five components: 1. An introduction to the brain, including a lesson on the concept of neuroplasticity, describing how and why our behaviors are controlled by thoughts and feelings in their brains, which have potential for change; 2. Written testimonials from older youths who describe their beliefs that people's personal traits (e.g., sadness, anxiety) are malleable, given the brain's plasticity; 3. Additional vignettes written by older youths, describing times when they used "growth mindsets" to persevere through social and emotional setbacks; 4. A summary of selected scientific studies suggesting that personality can, and often does, change in positive ways over time; and 5. An exercise in which the participants write notes to younger students, drawing on scientific information to describe the malleability of people's personal traits (i.e., a "self-persuasion" exercise).
  Arms: Project Personality
Behavioral: Sharing Feelings Intervention — The ST SSI is designed to control for nonspecific aspects of intervention, including engagement in a computer program. It includes the same number of reading and writing activities as the web-based growth mindset intervention; it also mirrors the web-based growth mindset intervention as closely as possible, including vignettes written by older youths who describe times when they benefited from sharing their feelings with friends or family.
  Arms: Sharing Feelings Intervention

SUMMARY:
Interventions for Autism Spectrum Disorder (ASD) are almost uniformly costly and time-intensive, blunting dissemination of intervention and stymying opportunities to make scalable impact. This study offers the first pilot randomized controlled trial (RCT) of whether a single session intervention, shown to reduce internalizing problems in typically-developing youth, may improve core and co-occuring symptoms of ASD.

DETAILED DESCRIPTION:
Interventions for core and co-occurring symptoms of autism spectrum disorders (ASD) are almost uniformly costly and time-intensive, blunting dissemination of intervention and stymying opportunities to make scalable, population-level impact. One promising solution to this problem is a new class of evidence-based treatments, single-session interventions (SSIs), which have shown remarkable efficacy in treating a range of other developmental psychopathologies. No study to date has examined SSIs in youth with ASD, which, if even marginally effective, could dramatically reduce the cost and expand the public health impact of accessible intervention options for ASD. This study offers the first pilot randomized controlled trial (RCT) of whether an SSI shown to reduce internalizing problems in typically-developing youth may improve core and co-occurring symptoms of ASD.

ELIGIBILITY:
Inclusion Criteria:

* Youth between the ages of 11-16 (inclusive) at the time of study participation;
* Youth with one parent or legal guardian willing to participate in the study (i.e. to be present for the lab visit and to complete questionnaires throughout the study period);
* Youth speaks English well enough to complete online or virtual based intervention activities;
* Youth with IQ ≥ 70;
* Parent or legal guardian speaks English well enough to complete online questionnaires;
* Youth with SCQ >10;
* Youth who meet criteria for autism or ASD on the ADOS-2.

Exclusion Criteria:

* Failure to meet the above inclusion criteria;
* Intellectual disability (IQ<70), as this may undermine comprehension of intervention materials;
* Adolescent is non-English speaking;
* The presence of a known developmental disability aside from ASD that would interfere with study participation;
* The presence of a significant medical disability or disorder that would interfere with study participation.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Children's Depression Inventory-2 (CDI-2) | up to 1 hour Pre-intervention
  Adolescent depressive symptom severity will be assessed using the Children's Depression Inventory-2 (CDI-2) Child and Parent forms. The CDI-2 is a reliable, valid measure of youth depression severity, normed for youth age and sex and yielding raw and T scores. Changes in youth CDI2 scores from baseline to each of the follow-up assessments will serve as the primary index of intervention effects. The CDI-2 will take approximately 15 minutes to complete. Each item on the child form is scored 0-2, yielding a total score between 0 and 56 with a higher total score indicating increased depressive symptomatology and a lower total score indicating decreased depressive symptomatology. Each item on the parent form is scored 0-3, yielding a total score between 0 and 51 with a higher score indicating increased depressive symptomatology and a lower total score indicating decreased depressive symptomatology.
Children's Depression Inventory-2 (CDI-2) | 3-moth followup
  Adolescent depressive symptom severity will be assessed using the Children's Depression Inventory-2 (CDI-2) Child and Parent forms. The CDI-2 is a reliable, valid measure of youth depression severity, normed for youth age and sex and yielding raw and T scores. Changes in youth CDI2 scores from baseline to each of the follow-up assessments will serve as the primary index of intervention effects. The CDI-2 will take approximately 15 minutes to complete. Each item on the child form is scored 0-2, yielding a total score between 0 and 56 with a higher total score indicating increased depressive symptomatology and a lower total score indicating decreased depressive symptomatology. Each item on the parent form is scored 0-3, yielding a total score between 0 and 51 with a higher score indicating increased depressive symptomatology and a lower total score indicating decreased depressive symptomatology.
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) | up to 1 hour Pre-intervention
  The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) is a valid, reliable tool for assessing executive functioning skills in home and school environments. Changes in BRIEF-2 scores from baseline to the 3-month follow-up assessment will serve as the primary index of intervention effects. The BRIEF-2 will take approximately 10 minutes. Each item on the child form is scored 1-3 (1 = Never; 2 = Sometimes; 3 = Often), yielding a total score between 55 and 165 with a higher total score indicating more severe deficiency. Each item on the parent form is scored 1-3 (1 = Never; 2 = Sometimes; 3 = Often), yielding a total scored between 55 and 165 with a higher total score indicating more severe deficiency.
Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) | 3-moth followup
  The Behavior Rating Inventory of Executive Function, Second Edition (BRIEF-2) is a valid, reliable tool for assessing executive functioning skills in home and school environments. Changes in BRIEF-2 scores from baseline to the 3-month follow-up assessment will serve as the primary index of intervention effects. The BRIEF-2 will take approximately 10 minutes. Each item on the child form is scored 1-3 (1 = Never; 2 = Sometimes; 3 = Often), yielding a total score between 55 and 165 with a higher total score indicating more severe deficiency. Each item on the parent form is scored 1-3 (1 = Never; 2 = Sometimes; 3 = Often), yielding a total scored between 55 and 165 with a higher total score indicating more severe deficiency.

SECONDARY OUTCOMES:
Brief Symptom Inventory 18 (BSI-18) | up to 1 hour Pre-intervention
  The Brief Symptom Inventory 18 (BSI-18) is a valid, reliable screening tool for adult (here, parental) psychological distress. Adult respondents rate endorsement of 18 physical and emotional complaints on a 0-4 Likert scale (0 = Not at all; 4 = Extremely), yielding a total between 0 and 72 with a higher score indicating increased parental stress. The BSI-18 includes 3 subscales for somatic, anxiety, and depressive symptoms, respectively. The total sum score yields an additional total distress score. The BSI-18 will take approximately 4 minutes to complete.
Brief Symptom Inventory 18 (BSI-18) | 3-month followup
  The Brief Symptom Inventory 18 (BSI-18) is a valid, reliable screening tool for adult (here, parental) psychological distress. Adult respondents rate endorsement of 18 physical and emotional complaints on a 0-4 Likert scale (0 = Not at all; 4 = Extremely), yielding a total between 0 and 72 with a higher score indicating increased parental stress. The BSI-18 includes 3 subscales for somatic, anxiety, and depressive symptoms, respectively. The total sum score yields an additional total distress score. The BSI-18 will take approximately 4 minutes to complete.
Multidimensional Anxiety Scale for Children-2 (MASC-2) | up to 1 hour Pre-intervention
  The Multidimensional Anxiety Scale for Children-2 (MASC-2) is widely-used in ASD studies. The parent- and self-report versions appear to measure the same construct in youths receiving the intervention and active control. It will be included in obtained models to see whether it alters patterns of effects. The MASC-2 will take approximately 15 minutes to complete. Each item is scored 0-3 (0 = Never; 3 = Often), yielding a total score between 0 and 150 with a higher total score indicating increased symptom severity.
Multidimensional Anxiety Scale for Children-2 (MASC-2) | 3-month followup
  The Multidimensional Anxiety Scale for Children-2 (MASC-2) is widely-used in ASD studies. The parent- and self-report versions appear to measure the same construct in youths receiving the intervention and active control. It will be included in obtained models to see whether it alters patterns of effects. The MASC-2 will take approximately 15 minutes to complete. Each item is scored 0-3 (0 = Never; 3 = Often), yielding a total score between 0 and 150 with a higher total score indicating increased symptom severity.
Primary Control Scale for Children (PCSC) | up to 1 hour Pre-intervention
  The Primary Control Scale for Children (PCSC) is a 24-item scale measuring youths' perceived ability to influence or alter objective events or conditions through personal effort. Youth rate agreement with statements about their ability to exert primary control (e.g., "I can do well on tests if I study hard"; "I can get other kids to like me if I try"). This PCSC has shown acceptable internal consistency, 6-month test-retest reliability, and strong inverse relations to adolescent depressive symptoms. The PCSC will take approximately 10 minutes to complete. Each item is scored 0-3, yielding a total score between 0 and 72, with an decreased total score indicating decreased ability to exert primary control.
Primary Control Scale for Children (PCSC) | up to 1 hour Post-intervention
  The Primary Control Scale for Children (PCSC) is a 24-item scale measuring youths' perceived ability to influence or alter objective events or conditions through personal effort. Youth rate agreement with statements about their ability to exert primary control (e.g., "I can do well on tests if I study hard"; "I can get other kids to like me if I try"). This PCSC has shown acceptable internal consistency, 6-month test-retest reliability, and strong inverse relations to adolescent depressive symptoms. The PCSC will take approximately 10 minutes to complete. Each item is scored 0-3, yielding a total score between 0 and 72, with an decreased total score indicating decreased ability to exert primary control.
Primary Control Scale for Children (PCSC) | 3-month followup
  The Primary Control Scale for Children (PCSC) is a 24-item scale measuring youths' perceived ability to influence or alter objective events or conditions through personal effort. Youth rate agreement with statements about their ability to exert primary control (e.g., "I can do well on tests if I study hard"; "I can get other kids to like me if I try"). This PCSC has shown acceptable internal consistency, 6-month test-retest reliability, and strong inverse relations to adolescent depressive symptoms. The PCSC will take approximately 10 minutes to complete. Each item is scored 0-3, yielding a total score between 0 and 72, with an decreased total score indicating decreased ability to exert primary control.
Secondary Control Scale for Children (SCSC) | up to 1 hour Pre-intervention
  The Secondary Control Scale for Children (SCSC) is a 20-item scale measuring youths' perceived ability to shape the personal impact of objective conditions on oneself, by adjusting oneself to fit those conditions. Youth rate agreement with items reflecting various kinds of secondary control, such as adjusting cognition ("When something bad happens, I can find a way to think about it that makes me feel better"). The SCSC has shown acceptable reliability and validity in a large youth sample. The SCSC will take approximately 5 minutes to complete. Each item is scored 0-3, yielding a total score between 0 and 60, with an decreased total score indicating decreased ability to exert primary control.
Secondary Control Scale for Children (SCSC) | up to 1 hour Post-intervention
  The Secondary Control Scale for Children (SCSC) is a 20-item scale measuring youths' perceived ability to shape the personal impact of objective conditions on oneself, by adjusting oneself to fit those conditions. Youth rate agreement with items reflecting various kinds of secondary control, such as adjusting cognition ("When something bad happens, I can find a way to think about it that makes me feel better"). The SCSC has shown acceptable reliability and validity in a large youth sample. The SCSC will take approximately 5 minutes to complete. Each item is scored 0-3, yielding a total score between 0 and 60, with an decreased total score indicating decreased ability to exert primary control.
Secondary Control Scale for Children (SCSC) | 3-month followup
  The Secondary Control Scale for Children (SCSC) is a 20-item scale measuring youths' perceived ability to shape the personal impact of objective conditions on oneself, by adjusting oneself to fit those conditions. Youth rate agreement with items reflecting various kinds of secondary control, such as adjusting cognition ("When something bad happens, I can find a way to think about it that makes me feel better"). The SCSC has shown acceptable reliability and validity in a large youth sample. The SCSC will take approximately 5 minutes to complete. Each item is scored 0-3, yielding a total score between 0 and 60, with an decreased total score indicating decreased ability to exert primary control.
Social Responsiveness Scale-2 (SRS-2) | up to 1 hour Pre-intervention
  The Social Responsiveness Scale-2 (SRS-2) is a 65-item scale measuring the parent's perceived presence, and severity, of current social deficits. Changes in the SRS-2 from baseline to the follow-up assessment will serve as the secondary index of intervention effects. The SRS-2 will take approximately 15 minutes to complete. Each item is scored 1-4, yielding a total score between 65 and 260 with a higher total score indicating increased deficiencies.
Social Responsiveness Scale-2 (SRS-2) | 3-moth followup
  The Social Responsiveness Scale-2 (SRS-2) is a 65-item scale measuring the parent's perceived presence, and severity, of current social deficits. Changes in the SRS-2 from baseline to the follow-up assessment will serve as the secondary index of intervention effects. The SRS-2 will take approximately 15 minutes to complete. Each item is scored 1-4, yielding a total score between 65 and 260 with a higher total score indicating increased deficiencies.
The Self Perception Profile for Children/ Adolescents (SPPC/A) self-report | up to 1 hour Pre-intervention
  The Self Perception Profile for Children/ Adolescents (SPPC/A) self-report is a short questionnaire that measures the self-esteem of youth. This measure will be administered in lab to parents and children. All SPPC/A will be administered by research assistants. The SPPC/A will take approximately 5 minutes to complete. Each item is scored 1-4, yielding a total score between 10 and 40 with a higher total score indicating increased social competence.
The Self Perception Profile for Children/ Adolescents (SPPC/A) self-report | up to 1 hour Post-intervention
  The Self Perception Profile for Children/ Adolescents (SPPC/A) self-report is a short questionnaire that measures the self-esteem of youth. This measure will be administered in lab to parents and children. All SPPC/A will be administered by research assistants. The SPPC/A will take approximately 5 minutes to complete. Each item is scored 1-4, yielding a total score between 10 and 40 with a higher total score indicating increased social competence.
The Self Perception Profile for Children/ Adolescents (SPPC/A) self-report | 3-month followup
  The Self Perception Profile for Children/ Adolescents (SPPC/A) self-report is a short questionnaire that measures the self-esteem of youth. This measure will be administered in lab to parents and children. All SPPC/A will be administered by research assistants. The SPPC/A will take approximately 5 minutes to complete. Each item is scored 1-4, yielding a total score between 10 and 40 with a higher total score indicating increased social competence.
Implicit Personality Theory Questionnaire (ITPQ) | up to 1 hour Pre-intervention
  The IPTQ asks youth to rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-7 Likert scale (e.g. "Your personality is something about you that you can't change very much"). Higher summed scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset. The ITPQ will take approximately 4 minutes to complete.
Implicit Personality Theory Questionnaire (ITPQ) | up to 1 hour Post-intervention
  The IPTQ asks youth to rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-7 Likert scale (e.g. "Your personality is something about you that you can't change very much"). Higher summed scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset. The ITPQ will take approximately 4 minutes to complete.
Implicit Personality Theory Questionnaire (ITPQ) | 3-month followup
  The IPTQ asks youth to rate the extent of their agreement with three statements linked to the malleability of personality, using a 1-to-7 Likert scale (e.g. "Your personality is something about you that you can't change very much"). Higher summed scores on these three items indicate a stronger fixed personality mindset, a lower scores, a stronger growth personality mindset. The ITPQ will take approximately 4 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Giacomantonio, B.S, Study Director — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buescher AV, Cidav Z, Knapp M, Mandell DS. Costs of autism spectrum disorders in the United Kingdom and the United States. JAMA Pediatr. 2014 Aug;168(8):721-8. doi: 10.1001/jamapediatrics.2014.210. PMID 24911948
- [Background] Kazdin AE, Blase SL. Rebooting Psychotherapy Research and Practice to Reduce the Burden of Mental Illness. Perspect Psychol Sci. 2011 Jan;6(1):21-37. doi: 10.1177/1745691610393527. Epub 2011 Feb 3. PMID 26162113
- [Background] Schleider JL, Weisz JR. Little Treatments, Promising Effects? Meta-Analysis of Single-Session Interventions for Youth Psychiatric Problems. J Am Acad Child Adolesc Psychiatry. 2017 Feb;56(2):107-115. doi: 10.1016/j.jaac.2016.11.007. Epub 2016 Nov 25. PMID 28117056
- [Background] Schleider J, Weisz J. A single-session growth mindset intervention for adolescent anxiety and depression: 9-month outcomes of a randomized trial. J Child Psychol Psychiatry. 2018 Feb;59(2):160-170. doi: 10.1111/jcpp.12811. Epub 2017 Sep 18. PMID 28921523
- [Background] Schleider JL, Weisz JR. Reducing risk for anxiety and depression in adolescents: Effects of a single-session intervention teaching that personality can change. Behav Res Ther. 2016 Dec;87:170-181. doi: 10.1016/j.brat.2016.09.011. Epub 2016 Sep 26. PMID 27697671
- [Background] Stice E, Burton E, Bearman SK, Rohde P. Randomized trial of a brief depression prevention program: an elusive search for a psychosocial placebo control condition. Behav Res Ther. 2007 May;45(5):863-76. doi: 10.1016/j.brat.2006.08.008. Epub 2006 Sep 27. PMID 17007812
- [Background] Aronson, E. (1999). The Power of Self-Persuasion. The American Psychologist, 54(11), 875-884. https://doi.org/10.1037/h0088188